CLINICAL TRIAL: NCT03335956
Title: A Double-blind, Randomised, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of SAD and MAD of CORT125281 in Healthy Subjects
Brief Title: CORT125281 Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CORT125281-600
Record Dates: First submitted 2017-10-31; First posted 2017-11-08 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Healthy
Keywords: Glucocorticoid receptor; antagonist
MeSH Terms: interventions — Prednisone; Pioglitazone; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (20):
- SAD Part 1 Placebo Cohort 1 Period 1 (Placebo Comparator)
  Interventions: Drug: Prednisone 25mg, fasted; Drug: Placebo oral capsule, fasted
- SAD Part 1 Active Cohort Period 1 (Experimental)
  Interventions: Drug: CORT125281, 40mg, fasted; Drug: Prednisone 25mg, fasted
- SAD Part 1 Placebo Cohort 1 Period 2 (Placebo Comparator)
  Interventions: Drug: Prednisone 25mg, fasted; Drug: Placebo oral capsule, fasted
- SAD Part 1 Active Cohort 1 Period 2 (Experimental)
  Interventions: Drug: Prednisone 25mg, fasted; Drug: CORT125281, 120mg, fasted
- SAD Part 1 Placebo Cohort 1 Period 3 (Placebo Comparator)
  Interventions: Drug: Prednisone 25mg, fasted; Drug: Placebo oral capsule, fasted
- SAD Part 1 Active Cohort 1 Period 3 (Experimental)
  Interventions: Drug: Prednisone 25mg, fasted; Drug: CORT125281, 360mg, fasted
- SAD Part 2 Placebo Cohort 2 Period 4 (Placebo Comparator)
  Interventions: Drug: Prednisone 25mg, fasted; Drug: Placebo oral capsule, fasted
- SAD Part 2 Active Cohort 2 Period 4 (Experimental)
  Interventions: Drug: Prednisone 25mg, fasted; Drug: CORT125281, 720mg, fasted
- SAD Part 2 Placebo Cohort 2 Period 5 (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule, fed; Drug: Prednisone 25mg, fed
- SAD Part 2 Active Cohort 2 Period 5 (Experimental)
  Interventions: Drug: Prednisone 25mg, fed; Drug: CORT125281, 360mg, fed
- SAD Part 2 Placebo Cohort 2 Period 6 (Placebo Comparator)
  Interventions: Drug: Prednisone 25mg, fasted; Drug: Placebo oral capsule
- SAD Part 2 Active Cohort 2 Period 6 (Experimental)
  Interventions: Drug: Prednisone 25mg, fasted; Drug: CORT125281, 360mg
- MAD Placebo Cohort 1 (Placebo Comparator)
  Interventions: Drug: Pioglitazone 15mg Tablet; Drug: Placebo oral capsule
- MAD Active Cohort 1 (Experimental)
  Interventions: Drug: Pioglitazone 15mg Tablet; Drug: CORT125281, 120mg
- MAD Placebo Cohort 2 (Placebo Comparator)
  Interventions: Drug: Pioglitazone 15mg Tablet; Drug: Placebo oral capsule
- MAD Active Cohort 2 (Experimental)
  Interventions: Drug: Pioglitazone 15mg Tablet; Drug: CORT125281, 180mg
- MAD Placebo Cohort 3 (Placebo Comparator)
  Interventions: Drug: Pioglitazone 15mg Tablet; Drug: Placebo oral capsule
- MAD Active Cohort 3 (Experimental)
  Interventions: Drug: Pioglitazone 15mg Tablet; Drug: CORT125281, 240mg
- MAD Placebo Cohort 4 (Placebo Comparator)
  Interventions: Drug: Pioglitazone 15mg Tablet; Drug: Placebo oral capsule
- MAD Active Cohort 4 (Experimental)
  Interventions: Drug: Pioglitazone 15mg Tablet; Drug: CORT125281, 360mg

INTERVENTIONS:
Drug: CORT125281, 40mg, fasted — CORT125281 is supplied as capsules for oral dosing
  Arms: SAD Part 1 Active Cohort Period 1
Drug: Prednisone 25mg, fasted — Challenge Agent, Dose and Route of Administration:
  Standard release 25 mg tablets, orally administered
  Arms: SAD Part 1 Active Cohort 1 Period 2; SAD Part 1 Active Cohort 1 Period 3; SAD Part 1 Active Cohort Period 1; SAD Part 1 Placebo Cohort 1 Period 1; SAD Part 1 Placebo Cohort 1 Period 2; SAD Part 1 Placebo Cohort 1 Period 3; SAD Part 2 Active Cohort 2 Period 4; SAD Part 2 Active Cohort 2 Period 6; SAD Part 2 Placebo Cohort 2 Period 4; SAD Part 2 Placebo Cohort 2 Period 6
Drug: Placebo oral capsule, fasted — Reference Therapy, Dose and Route of Administration:
  Placebo capsule, orally administered
  Arms: SAD Part 1 Placebo Cohort 1 Period 1; SAD Part 1 Placebo Cohort 1 Period 2; SAD Part 1 Placebo Cohort 1 Period 3; SAD Part 2 Placebo Cohort 2 Period 4
Drug: Pioglitazone 15mg Tablet — Probe Substrate, Dose and Route of Administration:
  15 Mg tablet, orally administered
  Arms: MAD Active Cohort 1; MAD Active Cohort 2; MAD Active Cohort 3; MAD Active Cohort 4; MAD Placebo Cohort 1; MAD Placebo Cohort 2; MAD Placebo Cohort 3; MAD Placebo Cohort 4
Drug: Placebo oral capsule, fed — Reference Therapy, Dose and Route of Administration:
  Placebo capsule, orally administered
  Arms: SAD Part 2 Placebo Cohort 2 Period 5
Drug: Prednisone 25mg, fed — Challenge Agent, Dose and Route of Administration:
  Standard release 25 mg tablets, orally administered
  Arms: SAD Part 2 Active Cohort 2 Period 5; SAD Part 2 Placebo Cohort 2 Period 5
Drug: CORT125281, 120mg, fasted — CORT125281 is supplied as capsules for oral dosing
  Arms: SAD Part 1 Active Cohort 1 Period 2
Drug: CORT125281, 360mg, fasted — CORT125281 is supplied as capsules for oral dosing
  Arms: SAD Part 1 Active Cohort 1 Period 3
Drug: CORT125281, 720mg, fasted — CORT125281 is supplied as capsules for oral dosing
  Arms: SAD Part 2 Active Cohort 2 Period 4
Drug: CORT125281, 360mg, fed — CORT125281 is supplied as capsules for oral dosing
  Arms: SAD Part 2 Active Cohort 2 Period 5
Drug: CORT125281, 360mg — CORT125281 is supplied as capsules for oral dosing twice, 12 hours apart, fasted (morning) and after evening meal
  Arms: SAD Part 2 Active Cohort 2 Period 6
Drug: CORT125281, 120mg — CORT125281 is supplied as capsules for oral dosing once daily
  Arms: MAD Active Cohort 1
Drug: CORT125281, 180mg — CORT125281 is supplied as capsules for oral dosing twice daily
  Arms: MAD Active Cohort 2
Drug: CORT125281, 240mg — CORT125281 is supplied as capsules for oral dosing twice daily
  Arms: MAD Active Cohort 3
Drug: CORT125281, 360mg — CORT125281 is supplied as capsules for oral dosing once daily
  Arms: MAD Active Cohort 4
Drug: Placebo oral capsule — Reference Therapy, Dose and Route of Administration:
  Placebo capsule, orally administered twice, 12 hours apart, fasted (morning) and after evening meal
  Arms: SAD Part 2 Placebo Cohort 2 Period 6
Drug: Placebo oral capsule — Reference Therapy, Dose and Route of Administration:
  Placebo capsule, orally administered, twice daily
  Arms: MAD Placebo Cohort 2; MAD Placebo Cohort 3
Drug: Placebo oral capsule — Reference Therapy, Dose and Route of Administration:
  Placebo capsule, orally administered, once daily
  Arms: MAD Placebo Cohort 1; MAD Placebo Cohort 4

SUMMARY:
This initial Phase I study will evaluate the dose-related safety and tolerability pharmacokinetics (PK) of CORT125281, and CORT125324 (active metabolite), and pharmacodynamics (PD) after single and multiple ascending oral doses of CORT125281 in healthy subjects.

DETAILED DESCRIPTION:
Separate single-and multiple-ascending dose (SAD and MAD) parts will be conducted. Throughout each part of the study, safety, pharmacological (PD) and PK effects will be assessed. Safety and tolerability will be assessed using adverse event (AE) monitoring, measurement of vital signs, recording 12-lead electrocardiogram (ECG), physical examination and clinical laboratory safety tests. Blood samples will be collected at intervals for assay of plasma concentration of CORT125281 and CORT125324.

The SAD part of the study is double-blind, randomized and placebo-controlled with respect to CORT125281. Two cohorts, each of 9 subjects, will receive three sequential single doses of the investigational medicinal product (IMP), either CORT125281 at the assigned dose level or placebo, in a partial within-subject crossover manner. The starting dose is CORT125281, 40 mg; the rules for determining later doses are detailed within the protocol. The PD effects of CORT125281 will be examined by testing its ability to ameliorate the pharmacological effects of a concomitantly administered dose of prednisone.

The MAD part of the study will be double-blind, randomized, placebo-controlled and parallel-group with respect to CORT125281. Up to four cohorts of 8 subjects, randomized so that 6 receive CORT125281 and 2 receive placebo, will participate in the study, so that up to four dose levels of CORT125281 are studied in total. An exploratory assessment will be made of the effect of repeated doses of CORT125281 on exposure to pioglitazone, probe substrate for CYP2C8. Each subject will be admitted on Day-1 for baseline assessments. On Day1, subjects will receive a single oral dose of pioglitazone, 15mg. From Day3 to Day16 (14 days), subjects will be dosed daily with IMP (CORT125281 at the selected dose or placebo). On Day13, subjects will receive a second dose of pioglitazone, 15 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Give written informed consent
2. If male, have undergone vasectomy, with no wish to have the procedure reversed
3. If female, using appropriate precautions to avoid pregnancy, defined as of nonchildbearing potential (ie, postmenopausal or permanently sterilised) or using highly effective contraception with low user-dependency

   * A woman is postmenopausal if it is more than 12 months since her last menstruation, without an alternative medical cause. A concentration of FSH in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy.
   * Accepted methods of permanent sterilization methods are hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
   * An IUD is the only acceptable method of highly effective contraception with low user-dependency, provided that the subject has tolerated its use for at least 3 months before the first dose of study medication and undertakes not to have it removed for 1 month after the last dose.
4. Be aged 18 to 65 years inclusive
5. Have a BMI of 19 to 30 kg/m2, inclusive
6. Be willing to comply with study restrictions as described in Section 4.6
7. Be able to comply with the requirements of the entire study
8. Be judged to be in good health, based upon the results of a medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory findings
9. For multiple dose cohorts, have a morning serum cortisol within the local reference range at screening and/or Day -1
10. Have suitable veins for multiple venepunctures/cannulation
11. Be able to swallow size 0 capsules whole

Exclusion Criteria:

1. Be an employee or immediate family member of the CRU or Corcept
2. Have been previously enrolled in this study
3. Have multiple drug allergies, or be allergic to any of the components of study medication, its matching placebo, challenge agents or probe substrates (see Section 5.1)
4. Have a condition that could be aggravated by glucocorticoid blockade (eg, asthma, any chronic inflammatory condition) or activation (eg, immunodeficiency, active infection) Subjects with inactive seasonal hay fever may be included. Subjects with childhood (aged less than 18 years) asthma may be included provided they have had no symptoms and required no treatment for at least 5 years
5. In the 6 calendar months before study drug administration, on average

   * Have smoked more than 5 cigarettes/day
   * Have consumed more than 14 units (female) or 21 units (male) of alcohol/week
   * Consumed liquorice or other glycyrrhetic acid derivatives regularly, in the judgement of the Investigator
6. In the 3 calendar months before study drug administration

   * Have donated blood or plasma in excess of 400 mL
   * Have participated in another clinical trial of a new chemical entity or a prescription medicine
7. Have a positive test for alcohol, smoking or drugs of abuse at screening or admission to any of the dosing sessions
8. Have clinically-relevant abnormal findings on vital signs, physical examination, laboratory screening tests, or 12-lead ECG, at screen and/or before first dose, including but not limited to:

   * Abnormal ECG waveform morphology that would preclude accurate measurement of the QT interval
   * QTcF >450 ms (from mean of 3 supine ECGs, performed at least 2 minutes apart)
   * Stage 2 or higher hypertension (supine/semi-recumbent systolic blood pressure [SBP] >160 mmHg; diastolic blood pressure [DBP] >100 mmHg, based on mean of duplicate values recorded at least 2 minutes apart)
   * Stage 1 hypertension (supine/semi-recumbent SBP 140-160 mmHg; DBP 90-100 mmHg, based on mean of duplicate values recorded at least 2 minutes apart) associated with indication for treatment ie, evidence of end-organ damage, diabetes or a 10 year cardiovascular risk, estimated using a standard calculator eg, QRisk2 2016 >20%
   * Glomerular filtration rate, estimated using the chronic kidney disease epidemiology (collaboration) (CKD-EPI) method (eGFR; see Section 6.2.5) <60 mL/minute/1.73 m2
   * Hypokalaemia (potassium below lower limit of normal)
   * ALT, AST and/or gammaglutamyl transferase (GGT) >1.5 times the upper limit of normal
   * Seropositive for hepatitis B, hepatitis C or human immunodeficiency viruses.
9. Have any medical or social reasons for not participating in the study raised by their General Practitioner/primary care physician
10. Have any other condition that might increase the risk to the individual or decrease the chance of obtaining satisfactory data, as assessed by the Investigator
11. Taken any prohibited prior medication, as described in Section 4.6.3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | SAD Cohorts Day 1 to Day 14; MAD Cohorts Day 1 to Day 30

SECONDARY OUTCOMES:
AUCtau Pharmacokinetic (PK) parameter | MAD Cohorts Day 3 to 19
  Area under the curve over a dose-interval (AUCtau)
AUC 0-tz PK parameter | CORT125281/CORT125324 - SAD Cohorts Day 1 to 4; MAD Cohorts Day 3 to 19; Pioglitizone - MAD Cohort Day 1 to 15
  Area under the curve from the time of dosing until the last quantifiable concentration (AUC 0-tz)
AUC 0-infinity PK parameter | CORT125281/CORT125324 - SAD Cohorts Day 1 to 4; MAD Cohorts Day 3 to 19; Pioglitizone - MAD Cohort Day 1 to 15
  Area under the curve from the time of dosing extrapolated to infinity (AUC 0-infinity)
Cmax PK parameter | CORT125281/CORT125324 - SAD Cohorts Day 1 to 4; MAD Cohorts Day 3 to 19; Pioglitizone - MAD Cohort Day 1 to 15
  Maximum concentration (Cmax)
Cmin PK parameter | MAD Cohorts Day 3 to 19
  Minimum concentration within a dose interval (Cmin)
Tmax PK parameter | SAD Cohorts Day 1 to 4; MAD Cohorts Day 3 to 19
  Time to maximum concentration (Tmax)
tlag PK parameter | SAD Cohorts Day 1 to 4; MAD Cohorts Day 3 to 19
  Latest time after dosing before the first quantifiable concentration (tlag)
apparent terminal rate constant PK parameter | SAD Cohorts Day 1 to 4; MAD Cohorts Day 3 to 19
t1/2 PK parameter | SAD Cohorts Day 1 to 4; MAD Cohorts Day 3 to 19
  Apparent terminal elimination half-life (t1/2)
MRT PK parameter | SAD Cohorts Day 1 to 4; MAD Cohorts Day 3 to 19
  Mean residence time (MRT)
Vz/F PK parameter | SAD Cohorts Day 1 to 4; MAD Cohorts Day 3 to 19
  Apparent oral volume of distribution during the terminal elimination phase (Vz/F)
CL/F PK parameter | SAD Cohorts Day 1 to 4; MAD Cohorts Day 3 to 19
  Apparent oral clearance (CL/F)
Observed accumulation ratio PK parameter | MAD Cohorts Day 3 to 19
4β-OH cholesterol PK parameter | MAD Cohorts Day 1 to Day 17
  4β-Hydroxycholesterol (4β-OH)
Pharmacodynamics (PD) Peripheral blood neutrophil, eosinophil and lymphocyte counts | SAD Cohorts pre-dose through 24 hours post dose
PD Serum osteocalcin | SAD Cohorts pre-dose through 24 hours post dose
PD Pre- and postprandial blood glucose | SAD Cohorts Day 1, pre-dose to 6 hours post dose
PD Cytokines | SAD Cohorts Day 1, pre-dose to 24 hours post dose; MAD Cohorts Day 3 to Day 10
PD T cell profiling by flow cytometry | SAD Cohorts Day 1, pre-dose to 24 hours post dose; MAD Cohorts Day 3 to Day 10
PD Gene expression for glucocorticoid-modulated genes | SAD Cohorts Day 1, pre-dose to 4 hours post dose
PD Cortisol | MAD Cohorts pre-dose to Day 16
PD ACTH | MAD Cohorts pre-dose to Day 16
  Adrenocorticotropic hormone (ACTH)
PD DHEA S | MAD Cohorts Day 3 to Day 16
  Dehydroepiandrosterone sulphate (DHEA-S)
PD androstenedione | MAD Cohorts Day 3 to Day 16
PD Fasting glucose | MAD Cohorts Day 1 to Day 13
PD insulin | MAD Cohorts Day 1 to Day 13
PD HOMA-IR | MAD Cohorts Day 1 to Day 13
  Homeostatic model assessment of insulin-resistance (HOMA-IR)

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Shepherd, M.D., Ph.D., Study Director — Corcept Therapeutics
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided